CLINICAL TRIAL: NCT02439463
Title: Traumatic Below-knee Amputees With Prosthetics: Health-related Quality of Life and Locomotor Capabilities
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, MD, Helsinki University Central Hospital
Other Study IDs: 364/13/03/02/2014/7
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Amputees

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Below-knee amputation — Patients with traumatic below-knee amputation.

SUMMARY:
The present study assesses the health-related quality of life and the locomotor capabilities major traumatic lower limb amputees who use prosthesis.

DETAILED DESCRIPTION:
A cross sectional study based on a retrospective review of prosthetic using major traumatic lower limb amputees' demographic and clinical details together with HRQoL and locomotor capabilities patient-reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Below-knee prosthesis users with amputation due to trauma
2. age >18

Exclusion Criteria:

1. Patients with no prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Below-knee amputees who use limb prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The health-related quality of life measured by HRQoL score | 2-5 years
Locomotor capabilities of traumatic below-knee amputees with prothesis | 2-5 years

SECONDARY OUTCOMES:
15D health-related quality of life instrument | 2-5 years
Prothesis Evaluation Questionnaire | 2-5 yeats

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J Tukiainen, MD,PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland